CLINICAL TRIAL: NCT07234578
Title: Analysis of Hip Rotator Strength and ROM in Amateur Soccer Players: A Cross-Sectional Study
Brief Title: Analysis of Hip Rotator Strength and ROM in Amateur Soccer Players
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Josep C. Benitez Martinez, Associate Professor, University of Valencia
Other Study IDs: 1662009173390
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hip Joint

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to analyze hip rotator strength and range of motion, comparing measurements taken with the hip positioned at 90° and 0°. Clinical history data, as well as hip strength and range of motion measurements, will be collected during the 2022/23 and 2023/24 seasons.

DETAILED DESCRIPTION:
This cross-sectional observational study aims to analyze the relationship between hip rotator strength and range of motion, comparing measurements taken with the hip positioned at 90° and at 0°. The study seeks to determine whether hip position influences the assessment of rotational strength and flexibility, providing useful information for both clinical evaluation and athletic performance monitoring. Data will be collected through direct measurements of hip strength and range of motion. Assessments will be performed during the 2022/23 and 2023/24 seasons. The findings are expected to contribute to a better understanding of how hip joint positioning affects rotator muscle function and mobility in healthy and active individuals.

ELIGIBILITY:
Inclusion Criteria:

* male amateur soccer players
* aged between 18-50
* players who were active participants in training sessions.

Exclusion Criteria:

* participants reporting current hip or groin pain, regardless of whether the pain resulted in time loss
* players with hip/groin injury in the preceding 4 months before study initiation
* players with longstanding injuries (>6 weeks) in the lower extremities
* previous injury or surgery in the lumbopelvic or hip region in the past year
* players with >2/10 on the Visual Analogue Scale during ROM and strength testing protocols of this study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Amateur soccer players from the Valencian region
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Hip Rotation Strength | At the time of assessment (single study visit)
  Maximal isometric strength of the hip internal and external rotator muscles measured at 0° and 90° of hip flexion.
Hip Rotation Range of Motion | At the time of assessment (single study visit)
  Passive range of motion for hip internal and external rotation measured at 0° and 90° of hip flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Benitez-Martinez, Dr, Principal Investigator — Universitat de Valencia
Locations (1):
- CD Serranos Valencia, Valencia, Valencia, Spain

REFERENCES:
- [Background] Hoglund LT, Wong AL, Rickards C. The impact of sagittal plane hip position on isometric force of hip external rotator and internal rotator muscles in healthy young adults. Int J Sports Phys Ther. 2014 Feb;9(1):58-67. PMID 24567856